CLINICAL TRIAL: NCT02773446
Title: Human Challenge Model Refinement for B7A, An Enterotoxigenic Escherichia Coli (ETEC) Challenge Strain That Expresses CS6
Brief Title: Human Challenge Model Refinement With Enterotoxigenic Escherichia Coli Strain B7A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); PATH (Other); Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CIR303 B7A
Record Dates: First submitted 2016-05-10; First posted 2016-05-16 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-04

CONDITIONS: Healthy Volunteer
Keywords: ETEC; Escherichia coli; enteritis; Challenge; CS6; Enterotoxigenic
MeSH Terms: conditions — Escherichia coli Infections; Enteritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 group A (Experimental): Volunteers will receive 8 logs of E. coli strain B7A after overnight fast
  Interventions: Biological: ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer
- Cohort 1 group B (Experimental): Volunteers will receive 9 logs of E. coli strain B7A after 90 minute fast
  Interventions: Biological: ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer
- Cohort 1 group C (Experimental): Volunteers will receive 9 logs of E. coli strain B7A after overnight fast
  Interventions: Biological: ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer
- Cohort 1 group D (Experimental): Volunteers will receive 10 logs of E. coli strain B7A after 90 minute fast
  Interventions: Biological: ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer
- Cohort 2 group A (Experimental): subjects from Cohort 1 who met primary endpoint will receive optimal regimen as determined by analysis after Cohort 1.
  Interventions: Biological: ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer
- Cohort 2 group B (Experimental): Naive subjects who will receive optimal regimen as determined by analysis after Cohort 1
  Interventions: Biological: ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer

INTERVENTIONS:
Biological: ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer — ETEC Bacteria

SUMMARY:
The purpose of this study is to determine the safe and optimal dose and regimen (fasting duration) for administering the challenge ETEC strain B7A, a CS6 expressing ETEC strain.

Additionally, an assessment of homologous protection following rechallenge with B7A will be assessed.

DETAILED DESCRIPTION:
Enterotoxigenic Escherichia coli (ETEC) is the most common causes of infectious diarrhea in children in resource limited countries, and is also a frequent cause of traveler's diarrhea in civilian and military travelers to endemic countries. ETEC strains express one or both of two enterotoxins (heat labile toxin (LT) and heat stable toxin (ST)) that cause help the bacteria cause the main symptom of watery diarrhea. They also express a variety of colonization factors (CF) that help them attach to the intestinal wall. Each colonization factor has one or more surface antigens (CS).

Vaccines and treatments to prevent ETEC disease are under development. Some of these target specific enterotoxins or colonization factors. For over 40 years, we have used ETEC human challenge studies to understand the ETEC disease process, immune response, and more recently, to determine whether treatments or vaccines are protective or effective in mitigating disease. One concern about these challenge study is the use of high doses of bacteria given may overwhelm the protective efficacy of the vaccine or treatment. Several strains of ETEC have been used in these challenge studies; a frequently used strain is B7A (CS6+, LT+, ST+. O148:H28).

This study will explore the optimal dosing strategy for B7A, in order to minimize the dose of ETEC necessary to produce disease in healthy adult volunteers. There will be two inpatient admissions. The first will examine 4 dosing and fasting regimens in healthy volunteers. The second admission will include volunteers who became ill during the first admission, as well as a new group of volunteers. This second admission will validate the optimal dose from the first admission, as well as to determine if previous infection with B7A ETEC will protect against a new infection. Trying to understand the immune response to this challenge organism may help us optimize vaccine design and delivery to protect people from this infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 50 years of age, inclusive.
2. General good health, without clinically significant medical history, physical examination findings or clinical laboratory abnormalities per clinical judgment of the PI.
3. Completion of a training session and demonstration of comprehension of the protocol procedures and knowledge of ETEC-associated illness by passing a written examination.
4. Willingness to participate after informed consent obtained.
5. Availability for the study duration, including all planned follow-up visits.
6. Negative pregnancy test with understanding to not become pregnant during the study or within three months following last scheduled study visit.

Exclusion Criteria:

1. Presence of a significant medical condition which in the opinion of the investigator precludes participation in the study.
2. Significant abnormalities in screening hematology or serum chemistry as determined by PI or PI in consultation with the research monitor and sponsor.
3. Evidence of confirmed infection with HIV, Hepatitis B, or Hepatitis C.
4. Evidence of Immunoglobulin A (IgA) deficiency (serum IgA < 7 mg/dL or below the limit of detection of assay).
5. Evidence of current excessive alcohol consumption or drug dependence (a targeted drug screen may be used to evaluate at the clinician's discretion).
6. Evidence of impaired immune function.
7. Recent vaccination or receipt of an investigational product (within 30 days before receipt of challenge).
8. Any other criteria which, in the investigator's opinion, would compromise the ability of the subject to participate in the study, the safety of the study, or the results of the study.
9. History of microbiologically confirmed ETEC or cholera infection in last 3 years.
10. Occupation involving handling of ETEC or Vibrio cholerae currently, or in the past 3 years.
11. Symptoms consistent with Travelers' Diarrhea concurrent with travel or planned travel to countries where ETEC infection is endemic.
12. Vaccination for or ingestion of ETEC, cholera, or E coli heat labile toxin within 3 years prior to dosing.
13. Any prior experimental infection with ETEC strain B7A.
14. Abnormal stool pattern.
15. Regular use of laxatives, antacids, or other agents to lower stomach acidity.
16. Use of any medication known to affect the immune function.
17. Known allergy to two of the following antibiotics: ciprofloxacin, trimethoprim-sulfamethoxazole, and amoxicillin.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar R. Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Center for Immunization Research, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be published in Peer reviewed journal

REFERENCES:
- [Background] Porter CK, Riddle MS, Alcala AN, Sack DA, Harro C, Chakraborty S, Gutierrez RL, Savarino SJ, Darsley M, McKenzie R, DeNearing B, Steinsland H, Tribble DR, Bourgeois AL. An Evidenced-Based Scale of Disease Severity following Human Challenge with Enteroxigenic Escherichia coli. PLoS One. 2016 Mar 3;11(3):e0149358. doi: 10.1371/journal.pone.0149358. eCollection 2016. PMID 26938983
- [Background] Harro C, Chakraborty S, Feller A, DeNearing B, Cage A, Ram M, Lundgren A, Svennerholm AM, Bourgeois AL, Walker RI, Sack DA. Refinement of a human challenge model for evaluation of enterotoxigenic Escherichia coli vaccines. Clin Vaccine Immunol. 2011 Oct;18(10):1719-27. doi: 10.1128/CVI.05194-11. Epub 2011 Aug 18. PMID 21852546
- [Background] Chakraborty S, Harro C, DeNearing B, Ram M, Feller A, Cage A, Bauers N, Bourgeois AL, Walker R, Sack DA. Characterization of Mucosal Immune Responses to Enterotoxigenic Escherichia coli Vaccine Antigens in a Human Challenge Model: Response Profiles after Primary Infection and Homologous Rechallenge with Strain H10407. Clin Vaccine Immunol. 2015 Nov 18;23(1):55-64. doi: 10.1128/CVI.00617-15. Print 2016 Jan. PMID 26581889
- [Background] Isidean SD, Riddle MS, Savarino SJ, Porter CK. A systematic review of ETEC epidemiology focusing on colonization factor and toxin expression. Vaccine. 2011 Aug 26;29(37):6167-78. doi: 10.1016/j.vaccine.2011.06.084. Epub 2011 Jul 1. PMID 21723899
- [Background] Ahmed T, Bhuiyan TR, Zaman K, Sinclair D, Qadri F. Vaccines for preventing enterotoxigenic Escherichia coli (ETEC) diarrhoea. Cochrane Database Syst Rev. 2013 Jul 5;2013(7):CD009029. doi: 10.1002/14651858.CD009029.pub2. PMID 23828581
- [Background] McKenzie R, Porter CK, Cantrell JA, Denearing B, O'Dowd A, Grahek SL, Sincock SA, Woods C, Sebeny P, Sack DA, Tribble DR, Bourgeois AL, Savarino SJ. Volunteer challenge with enterotoxigenic Escherichia coli that express intestinal colonization factor fimbriae CS17 and CS19. J Infect Dis. 2011 Jul 1;204(1):60-4. doi: 10.1093/infdis/jir220. PMID 21628659
- [Background] Porter CK, Riddle MS, Tribble DR, Louis Bougeois A, McKenzie R, Isidean SD, Sebeny P, Savarino SJ. A systematic review of experimental infections with enterotoxigenic Escherichia coli (ETEC). Vaccine. 2011 Aug 11;29(35):5869-85. doi: 10.1016/j.vaccine.2011.05.021. Epub 2011 May 25. PMID 21616116
- [Background] Lamberti LM, Bourgeois AL, Fischer Walker CL, Black RE, Sack D. Estimating diarrheal illness and deaths attributable to Shigellae and enterotoxigenic Escherichia coli among older children, adolescents, and adults in South Asia and Africa. PLoS Negl Trop Dis. 2014 Feb 13;8(2):e2705. doi: 10.1371/journal.pntd.0002705. eCollection 2014 Feb. PMID 24551265
- [Background] Lanata CF, Fischer-Walker CL, Olascoaga AC, Torres CX, Aryee MJ, Black RE; Child Health Epidemiology Reference Group of the World Health Organization and UNICEF. Global causes of diarrheal disease mortality in children <5 years of age: a systematic review. PLoS One. 2013 Sep 4;8(9):e72788. doi: 10.1371/journal.pone.0072788. eCollection 2013. PMID 24023773

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohort 2 group A consists of 11 subjects from Cohort 1. These subjects were re admitted for a second admission. The total number of subjects enrolled was 47.
Period: First Admission
Arm/Group | Cohort 1 Group A | Cohort 1 Group B | Cohort 1 Group C | Cohort 1 Group D | Cohort 2 Group A | Cohort 2 Group B
Started | 7 | 7 | 7 | 7 | 0 | 0
Completed | 6 | 7 | 7 | 6 | 0 | 0
Not Completed | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Period: Second Admission
Arm/Group | Cohort 1 Group A | Cohort 1 Group B | Cohort 1 Group C | Cohort 1 Group D | Cohort 2 Group A | Cohort 2 Group B
Started | 0 | 0 | 0 | 0 | 11 | 19
Completed | 0 | 0 | 0 | 0 | 11 | 19
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cohort 2 group A consists of 11 subjects from Cohort 1. These subjects were re admitted for a second admission. The total number of subjects enrolled was 47.
Groups:
- Cohort 1 Group A: 8 logs of E. coli strain B7A after overnight fast
  ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer: ETEC Bacteria
- Cohort 1 Group B: 9 logs of E. coli strain B7A after 90 minute fast
  ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer: ETEC Bacteria
- Cohort 1 Group C: 9 logs of E. coli strain B7A after overnight fast
  ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer: ETEC Bacteria
- Cohort 1 Group D: 10 logs of E. coli strain B7A after 90 minute fast
  ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer: ETEC Bacteria
- Cohort 2 Group A: subjects from Cohort 1 who met primary endpoint - 9 logs of E.coli strain B7A
  ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer: ETEC Bacteria
- Cohort 2 Group B: Naive subjects - 9 logs of E. coli strain B7A after overnight fast
  ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer: ETEC Bacteria
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Group A | Cohort 1 Group B | Cohort 1 Group C | Cohort 1 Group D | Cohort 2 Group A | Cohort 2 Group B | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 11 | 19 | 58
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Cohort 2 group A consists of 11 subjects from Cohort 1. These subjects were re admitted for a second admission. The total number of subjects enrolled was 47. Each cohort was analyzed separately.
  years
    Cohort 1: number analyzed (Participants) | 7 | 7 | 7 | 7 | 0 | 0 | 28
    Cohort 1 | 36 [29.5 to 39] | 34 [31.5 to 37] | 39 [31 to 40.5] | 35 [33 to 40.5] |  |  | 34.5 [32 to 40]
    Cohort 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 19 | 30
    Cohort 2 |  |  |  |  | 39 [32 to 41] | 35 [30 to 42] | 36 [30 to 41.5]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Cohort 2 group A consists of 11 subjects from Cohort 1. These subjects were re admitted for a second admission. The total number of subjects enrolled was 47. Each cohort was analyzed separately.
  Participants
    Cohort 1: number analyzed (Participants) | 7 | 7 | 7 | 7 | 0 | 0 | 28
    Cohort 1: Female | 2 | 3 | 2 | 1 | 0 | 0 | 8
    Cohort 1: Male | 5 | 4 | 5 | 6 | 0 | 0 | 20
    Cohort 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 19 | 30
    Cohort 2: Female | 0 | 0 | 0 | 0 | 3 | 5 | 8
    Cohort 2: Male | 0 | 0 | 0 | 0 | 8 | 14 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Cohort 2 group A consists of 11 subjects from Cohort 1. These subjects were re admitted for a second admission. The total number of subjects enrolled was 47. Each cohort was analyzed separately.
  Participants
    Cohort 1: number analyzed (Participants) | 7 | 7 | 7 | 7 | 0 | 0 | 28
    Cohort 1: Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Cohort 1: Not Hispanic or Latino | 7 | 6 | 7 | 7 | 0 | 0 | 27
    Cohort 1: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Cohort 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 19 | 30
    Cohort 2: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 5 | 5
    Cohort 2: Not Hispanic or Latino | 0 | 0 | 0 | 0 | 11 | 14 | 25
    Cohort 2: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Cohort 2 group A consists of 11 subjects from Cohort 1. These subjects were re admitted for a second admission. The total number of subjects enrolled was 47. Each cohort was analyzed separately.
  Participants
    Cohort 1: number analyzed (Participants) | 7 | 7 | 7 | 7 | 0 | 0 | 28
    Cohort 1: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Cohort 1: Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Cohort 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Cohort 1: Black or African American | 5 | 6 | 7 | 6 | 0 | 0 | 24
    Cohort 1: White | 1 | 1 | 0 | 1 | 0 | 0 | 3
    Cohort 1: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Cohort 1: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Cohort 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 19 | 30
    Cohort 2: American Indian or Alaska Native |  |  |  |  | 0 | 0 | 0
    Cohort 2: Asian |  |  |  |  | 0 | 1 | 1
    Cohort 2: Native Hawaiian or Other Pacific Islander |  |  |  |  | 0 | 0 | 0
    Cohort 2: Black or African American |  |  |  |  | 11 | 13 | 24
    Cohort 2: White |  |  |  |  | 0 | 2 | 2
    Cohort 2: More than one race |  |  |  |  | 0 | 0 | 0
    Cohort 2: Unknown or Not Reported |  |  |  |  | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Cohort 1 | 7 | 7 | 7 | 7 | 0 | 0 | 28
  United States: Cohort 2 | 0 | 0 | 0 | 0 | 11 | 19 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Safety- Solicited Symptoms Related to Challenge Administration
Description: Solicited symptoms (vomiting, abdominal pain, bloating, lightheadedness, anorexia, generalized myalgia, arthralgias, abdominal cramping, constipation, nausea, malaise, headache, flatulence)
Time Frame: 6 days post-challenge
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2 Group A: subjects from Cohort 1 who met primary endpoint 9 logs of E.coli strain B7A after overnight fast
  ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer: ETEC Bacteria
Arm/Group | Cohort 1 Group A | Cohort 1 Group B | Cohort 1 Group C | Cohort 1 Group D | Cohort 2 Group A | Cohort 2 Group B
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 11 | 19
Participants
  Vomiting | 0 | 0 | 3 | 2 | 1 | 3
  Abdominal Pain | 3 | 4 | 5 | 4 | 7 | 12
  Bloating | 5 | 6 | 5 | 4 | 5 | 11
  Lightheadedness | 1 | 4 | 4 | 1 | 2 | 3
  Anorexia | 4 | 4 | 5 | 4 | 4 | 14
  Generalized Myalgia | 0 | 1 | 0 | 1 | 2 | 3
  Arthralgias | 0 | 1 | 0 | 1 | 1 | 3
  Abdominal Cramping | 5 | 5 | 5 | 3 | 7 | 13
  Constipation | 1 | 1 | 2 | 0 | 0 | 0
  Nausea | 3 | 3 | 4 | 3 | 3 | 8
  Malaise | 4 | 4 | 4 | 3 | 4 | 10
  Headache | 3 | 4 | 4 | 5 | 4 | 10
  Flatulence | 7 | 6 | 6 | 4 | 7 | 10

2. Primary Outcome: Moderate-severe Diarrhea
Description: Moderate-severe diarrhea post challenge defined as
  * moderate diarrhea: 4 to 5 loose/liquid stools or 401-800 of loose/liquid stool in any 24-hour period
  * Severe diarrhea greater than or equal to 6 loose/liquid stools or greater than 800 g of loose/liquid stools in any 24-hour period
Time Frame: 5 days post challenge (Cohort 1 and Cohort 2 group B) 7 days post challenge (Cohort 2 Group A)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2 Group A: subjects from Cohort 1 who met primary endpoint- 9 logs of E. coli strain B7A after overnight fast
- Cohort 2 Group B: Naive subjects -9 logs of E. coli strain B7A after overnight fast
  ETEC strain B7A (O148:H28 CS6+ LT+ST+) (Lot 0481) in Buffer: ETEC Bacteria
Arm/Group | Cohort 1 Group A | Cohort 1 Group B | Cohort 1 Group C | Cohort 1 Group D | Cohort 2 Group A | Cohort 2 Group B
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 11 | 19
Participants | 3 | 3 | 5 | 5 | 5 | 11

3. Primary Outcome: Moderate-severe Diarrhea in Subjects Receiving Homologous Rechallenge
Description: Moderate-severe diarrhea post-challenge defined as
  * Moderate diarrhea: 4 to 5 loose/liquid stools or 401-800g of loose/liquid stool in any 24- hour period
  * Severe diarrhea: greater than or equal to 6 loose/liquid stools or greater than 800 g of loose/liquid stool in any 24-hour period
Time Frame: 7 days post-challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 Group A
Number analyzed (Participants) | 11
Participants | 5

4. Primary Outcome: Number of Participants With Safety -Solicited Symptoms Unrelated to Challenge Administration
Description: Safety solicited symptoms unrelated to challenge administration (vomiting, abdominal pain, bloating, lightheadedness, anorexia, generalized myalgia, arthralgias, abdominal cramping, constipation, nausea, malaise, headache, flatulence)
Time Frame: 6 days post-challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Group A | Cohort 1 Group B | Cohort 1 Group C | Cohort 1 Group D | Cohort 2 Group A | Cohort 2 Group B
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 11 | 19
Participants
  Vomiting | 1 | 0 | 0 | 0 | 0 | 0
  Abdominal pain | 0 | 0 | 0 | 0 | 0 | 0
  Bloating | 0 | 0 | 0 | 0 | 0 | 0
  Lightheadedness | 0 | 0 | 0 | 0 | 0 | 0
  Anorexia | 1 | 1 | 0 | 0 | 0 | 0
  Generalized myalgia | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgias | 0 | 0 | 0 | 0 | 1 | 0
  Abdominal Cramping | 0 | 0 | 0 | 0 | 0 | 0
  Constipation | 0 | 0 | 0 | 0 | 0 | 0
  Nausea | 1 | 0 | 0 | 0 | 0 | 0
  Malaise | 1 | 0 | 0 | 0 | 0 | 0
  Headache | 1 | 1 | 1 | 0 | 0 | 0
  Flatulence | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Immune Response to Challenge (Serology)
Time Frame: 28 days post challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Group A | Cohort 1 Group B | Cohort 1 Group C | Cohort 1 Group D | Cohort 2 Group A | Cohort 2 Group B
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 11 | 19
Participants
  IgG C66 | 1 | 3 | 0 | 0 | 3 | 4
  IgG LT | 2 | 1 | 3 | 4 | 6 | 10
  IgG LPS | 2 | 2 | 1 | 4 | 4 | 7
  IgA CS6 | 1 | 1 | 2 | 0 | 1 | 2
  IgA LT | 1 | 0 | 2 | 1 | 4 | 3
  IgA LPS | 5 | 6 | 4 | 7 | 6 | 18

6. Secondary Outcome: Immune Response to Challenge
Description: Antibody in Lymphocyte Supernatant (ALS) Immunoglobin G (IgG) (CS6) coli surface antigen 6 Immunoglobin G (IgG) heat labile Toxin (LT) Immunoglobin G (IgG) (LPS) Lipopolysaccharide Immunoglobin A (IgA) (CS6) coli surface antigen 6 Immunoglobin A (IgA) heat labile Toxin (LT) Immunoglobin A (IgG) (LPS) Lipopolysaccharide
Time Frame: 6 days post challenge
Population: samples for ALS IgG and IgA were unavailable for 1 participant in cohort 2 group A Samples for ALS IgG CS6, LT and IgA CS6 were unavailable for 1 participant in cohort 2 group B
Measure: Number; unit: participants
Arm/Group | Cohort 1 Group A | Cohort 1 Group B | Cohort 1 Group C | Cohort 1 Group D | Cohort 2 Group A | Cohort 2 Group B
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 11 | 19
participants
  IgG C66: number analyzed (Participants) | 7 | 7 | 7 | 7 | 10 | 18
  IgG C66 | 2 | 2 | 0 | 1 | 5 | 6
  IgG LT: number analyzed (Participants) | 7 | 7 | 7 | 7 | 10 | 18
  IgG LT | 1 | 2 | 4 | 2 | 8 | 9
  IgG LPS: number analyzed (Participants) | 7 | 7 | 7 | 7 | 10 | 19
  IgG LPS | 3 | 3 | 1 | 5 | 3 | 18
  IgA CS6: number analyzed (Participants) | 7 | 7 | 7 | 7 | 10 | 18
  IgA CS6 | 3 | 4 | 0 | 2 | 6 | 6
  IgA LT: number analyzed (Participants) | 7 | 7 | 7 | 7 | 10 | 19
  IgA LT | 1 | 0 | 1 | 1 | 4 | 8
  IgA LPS: number analyzed (Participants) | 7 | 7 | 7 | 7 | 10 | 19
  IgA LPS | 5 | 7 | 5 | 6 | 8 | 19

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Cohort 1 Group A | Cohort 1 Group B | Cohort 1 Group C | Cohort 1 Group D | Cohort 2 Group A | Cohort 2 Group B
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7 | 0/11 | 1/19
Other Adverse Events (participants affected / at risk) | 5/7 | 3/7 | 7/7 | 3/7 | 4/11 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Group A (N=7) | Cohort 1 Group B (N=7) | Cohort 1 Group C (N=7) | Cohort 1 Group D (N=7) | Cohort 2 Group A (N=11) | Cohort 2 Group B (N=19)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (19)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Group A (N=7) | Cohort 1 Group B (N=7) | Cohort 1 Group C (N=7) | Cohort 1 Group D (N=7) | Cohort 2 Group A (N=11) | Cohort 2 Group B (N=19)
Abdominal Distention (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
High pitched bowel sounds (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperactive Bowel Sounds (Gastrointestinal disorders) | 5 (5) | 2 (2) | 7 (7) | 3 (3) | 3 (3) | 8 (8)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypovolemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No